CLINICAL TRIAL: NCT04665765
Title: A Phase 2 Study of Polatuzumab Vedotin With Rituximab, Ifosfamide, Carboplatin, and Etoposide (PolaR-ICE) as Initial Salvage Therapy for Relapsed/Refractory Diffuse Large B-cell Lymphoma
Brief Title: Polatuzumab Vedotin, Rituximab, Ifosfamide, Carboplatin, and Etoposide (PolaR-ICE) as Initial Salvage Therapy for the Treatment of Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20148; NCI-2020-08524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20148 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-Cell Lymphoma Unclassifiable; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Primary Mediastinal (Thymic) Large B-Cell Cell Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Carboplatin; Etoposide; Ifosfamide; polatuzumab vedotin; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PolaR-ICE) (Experimental): SALVAGE THERAPY: Patients receive polatuzumab vedotin IV on day 1, rituximab IV on day 1, etoposide IV on days 1-3, carboplatin IV on day 2, and ifosfamide IV on day 2 or days 1-3. Treatment repeats every 21 days for up to 2-3 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response or stable disease by C2D15 may receive 1 additional cycle of PolaR-ICE IV.
  CONSOLIDATION THERAPY: Within 30-60 days after ASCT, patients receive polatuzumab vedotin IV on day 1. Treatment repeats every 21 days for up to 3-4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Ifosfamide; Drug: Polatuzumab Vedotin; Biological: Rituximab

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Drug: Polatuzumab Vedotin — Given IV
  Other Names: ADC DCDS4501A; Antibody-Drug Conjugate DCDS4501A; DCDS4501A; FCU 2711; polatuzumab vedotin-piiq; Polivy; RG7596; Ro 5541077-000
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase II trial studies the effect of polatuzumab vedotin, rituximab, ifosfamide, carboplatin, and etoposide as initial salvage therapy in treating patients with diffuse large B-cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Polatuzumab vedotin is a monoclonal antibody, polatuzumab, linked to a toxic agent called vedotin. Polatuzumab attaches to CD79b positive cancer cells in a targeted way and delivers vedotin to kill them. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Chemotherapy drugs, such as ifosfamide, carboplatin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy with immunotherapy may kill more cancer cells in patients with diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety and tolerability of polatuzumab vedotin (Pola) added to rituximab, ifosfamide, carboplatin, and etoposide (PolaR-ICE) as first salvage therapy for relapsed or refractory (R/R) diffuse large B-cell lymphoma (DLBCL). (Safety Lead-in) II. Evaluate the anti-tumor activity of PolaR-ICE as first salvage therapy for R/R DLBCL as assessed by the complete response rate after 2 cycles. (Phase 2)

SECONDARY OBJECTIVES:

I. Evaluate the overall response rate to PolaR-ICE as first salvage therapy for R/R DLBCL.

II. Evaluate the progression-free and overall survival of patients who received PolaR-ICE as first salvage therapy for R/R DLBCL followed by autologous stem cell transplantation (ASCT) and single-agent Pola consolidation after ASCT.

III. Evaluate the CR rate after Pola consolidation among those who were partial response (PR) at ASCT.

IV. Evaluate the toxicity of PolaR-ICE salvage therapy and that of Pola consolidation after ASCT.

V. Assess the rate of stem cell mobilization and collection failure in patients with R/R DLBCL who receive PolaR-ICE as first salvage therapy.

EXPLORATORY OBJECTIVES:

I. Assess the kinetics of circulating tumor deoxyribonucleic acid (DNA) after PolaR-ICE as first salvage therapy for R/R DLBCL followed by ASCT and single-agent Pola consolidation after ASCT.

II. Assess possible biomarkers of response to PolaR-ICE in patients with R/R DLBCL.

III. Examine the association between clinical outcomes (response, progression-free survival [PFS]) and pathological tumor characteristics.

IV. Examine the association between clinical outcomes (response, PFS) and circulating tumor (ct)DNA characteristics (mutation profile, kinetics of clearance).

OUTLINE:

SALVAGE THERAPY: Patients receive polatuzumab vedotin intravenously (IV) on day 1, rituximab IV on day 1, etoposide IV on days 1-3, carboplatin IV on day 2, and ifosfamide IV on day 2 or days 1-3. Treatment repeats every 21 days for up to 2-3 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response or stable disease by cycle 2 day 15 (C2D15) may receive 1 additional cycle of PolaR-ICE IV.

CONSOLIDATION THERAPY: Within 30-60 days after ASCT, patients receive polatuzumab vedotin IV on day 1. Treatment repeats every 21 days for up to 3-4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, and then periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Be willing to provide archival tissue of a biopsy that was performed after the frontline systemic therapy

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Histologically confirmed diagnosis of diffuse large B-cell lymphoma according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution. Subtypes of DLBCL including transformed indolent lymphomas (TIL), primary mediastinal large B-cell lymphoma (PMBCL), and aggressive B-cell lymphoma unclassified (BCL-U) are eligible
* Biopsy-proven relapsed or refractory disease after 1 line of frontline CD20-directed immunotherapy with anthracycline- or anthracenedione-based multi-agent chemotherapy. Monotherapy with rituximab or other CD20-directed immunotherapy prior to frontline chemotherapy or as maintenance therapy, and radiation therapy in a limited field or as a part of the frontline treatment plan are permitted
* Prior lymphoma therapy should be completed at least 2 weeks before start of protocol therapy
* Measurable disease by computed tomography (CT) or positron emission tomography (PET)/CT scan with one or more sites of disease >= 1.5 cm in longest dimension
* Considered eligible for high-dose chemotherapy followed by ASCT
* Fully recovered from the acute toxic effects (except alopecia) to =< grade 1 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) >= 1,000/mm^3 (without bone marrow involvement)

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* ANC >= 750/mm^3 (with bone marrow involvement)

  * NOTE: Growth factor is not permitted within 7 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 100,000/mm^3 (without bone marrow involvement)

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Platelets >= 75,000/mm^3 (with bone marrow involvement)

  * NOTE: Platelet transfusions are not permitted within 7 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin >= 8 g/dL (no erythropoietin and/or packed red blood cells (pRBC) transfusion allowed within 7 days prior to screening)
* Total bilirubin =< 1.5 X upper limit of normal (ULN). If hepatic involvement by lymphoma, or Gilbert's disease: =< 3 X ULN
* Aspartate aminotransferase (AST) =< 2.5 x ULN. If hepatic involvement by lymphoma: AST =< 5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN. If hepatic involvement by lymphoma: ALT =< 5 x ULN
* Creatinine clearance of >= 50 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: international normalized ratio (INR) OR prothrombin (prothrombin time [PT]) =< 1.5 x ULN. If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: activated partial thromboplastin time (aPTT) =< 1.5 x ULN. If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 12 months after the last dose of polatuzumab vedotin or rituximab for women, at least 5 months following the last dose of polatuzumab vedotin or 3 months following the last dose of rituximab for men, and at least 6 months following the last dose of ifosfamide, carboplatin, or etoposide for both women and men

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Patients who are not hematopoietic stem cell transplant candidates are excluded
* Prior solid organ transplantation
* Systemic steroid therapy or any other form of immunosuppressive therapy for lymphoma symptom control must be tapered down to =< 10 mg/day prednisone or equivalent. Exceptions are:

  * Inhaled or topical steroids
  * Adrenal replacement doses > 10 mg daily prednisone equivalents in the absence of active autoimmune disease
* Peripheral neuropathy >= grade 2 or demyelinating form of Charcot-Marie-Tooth disease
* Known active central nervous system (CNS) involvement by lymphoma, including leptomeningeal involvement
* Active infection requiring systemic therapy
* Other active malignancy requiring therapy. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to study agents
* Recent major surgery (within 4 weeks) prior to start of protocol therapy, other than for diagnosis
* Symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias), cerebrovascular event/stroke or myocardial infarction within the past 6 months
* Known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. Patients with past HBV infection (defined as negative hepatitis B surface antigen [HBsAg] and positive hepatitis B core antibody [HBcAb]) are eligible if HBV DNA is undetectable. Patients who are positive for HCV antibody are eligible if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA). Testing to be done only in patients suspected of having infections or exposures
* Known active human immunodeficiency virus (HIV) infection. Subjects who have an undetectable or unquantifiable HIV viral load with CD4 >= 200 and are on highly active antiretroviral therapy (HAART) medication are allowed. Testing to be done only in patients suspected of having infections or exposures
* History of or current progressive multifocal leukoencephalopathy (PML)
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2026-07-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex F Herrera, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Emory University, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Safety Lead-In; Phase II: SALVAGE THERAPY: Patients receive polatuzumab vedotin IV on day 1, rituximab IV on day 1, etoposide IV on days 1-3, carboplatin IV on day 2, and ifosfamide IV on day 2 or days 1-3. Treatment repeats every 21 days for up to 2-3 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response or stable disease by C2D15 may receive 1 additional cycle of PolaR-ICE IV.
  CONSOLIDATION THERAPY: Within 30-60 days after ASCT, patients receive polatuzumab vedotin IV on day 1. Treatment repeats every 21 days for up to 3-4 cycles in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Polatuzumab Vedotin: Given IV
  Rituximab: Given IV
Period: Overall Study
Arm/Group | Safety Lead-In | Phase II
Started | 6 | 35
Completed | 6 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-In | Phase II | Total
Number analyzed (Participants) | 6 | 35 | 41
Age, Continuous [Median (Full Range); unit: years] | 57 [34 to 75] | 65 [21 to 81] | 65 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 3 | 24 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 3 | 29 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 4 | 28 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 35 | 41
Histology at On-Study [Count of Participants; unit: Participants]
  Diffuse large B cell lymphoma NOS/De Novo | 4 | 23 | 27
  Transformed Lymphoma | 2 | 9 | 11
  Primary mediastinal large B cell lymphoma | 0 | 3 | 3
B Symptoms at On-Study [Count of Participants; unit: Participants]
  B Symptoms | 1 | 7 | 8
  Absence of B symptoms | 5 | 28 | 33

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate After Two Cycles of PolaR-ICE Salvage Therapy
Description: Estimated by the proportion of response-evaluable patients achieving CR after 2 cycles of salvage therapy, along with the 95% exact binomial confidence interval. Polatuzumab vedotin (Pola) was added to rituximab, ifosfamide, carboplatin, and etoposide (PolaR-ICE) as salvage therapy.
Time Frame: After 2 cycles of salvage therapy (each cycle is 21 days)
Population: Three subjects in Phase II were not evaluable for they did not finish two cycles of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Lead-In | Phase II
Number analyzed (Participants) | 6 | 32
percentage of participants | 67 [22 to 96] | 59 [41 to 76]

2. Primary Outcome: Number of Unacceptable Toxicities of PolaR-ICE Salvage Therapy (Phase 2 Stage)
Description: Unacceptable toxicity was defined as the events in Section 11.2 occurring during the first 2 cycles of treatment that was at least possibly related to study treatment.
Time Frame: During the first 2 cycles of PolaR-ICE salvage therapy (each cycle is 21 days)
Measure: Number; unit: events
Groups:
- Treatment (PolaR-ICE): SALVAGE THERAPY: Patients receive polatuzumab vedotin IV on day 1, rituximab IV on day 1, etoposide IV on days 1-3, carboplatin IV on day 2, and ifosfamide IV on day 2 or days 1-3. Treatment repeats every 21 days for up to 2-3 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response or stable disease by C2D15 may receive 1 additional cycle of PolaR-ICE IV.
  CONSOLIDATION THERAPY: Within 30-60 days after ASCT, patients receive polatuzumab vedotin IV on day 1. Treatment repeats every 21 days for up to 3-4 cycles in the absence of disease progression or unacceptable toxicity.
  Carboplatin: Given IV
  Etoposide: Given IV
  Ifosfamide: Given IV
  Polatuzumab Vedotin: Given IV
  Rituximab: Given IV
Arm/Group | Treatment (PolaR-ICE)
Number analyzed (Participants) | 35
events | 0

3. Primary Outcome: Number of Unacceptable Toxicities of PolaR-ICE Salvage Therapy (Safety lead-in Stage)
Description: as for outcome 2
Time Frame: During the first 2 cycles of PolaR-ICE salvage therapy (each cycle is 21 days)
Measure: Number; unit: events
Arm/Group | Treatment (PolaR-ICE)
Number analyzed (Participants) | 5
events | 0

4. Secondary Outcome: Overall Response Rate (ORR) of the PolaR-ICE Salvage Therapy
Description: Estimated by the proportion of response-evaluable participants that achieve a best response of either CR or partial response (PR) at the end of PolaR-ICE therapy, along with the 95% exact binomial confidence interval. Polatuzumab vedotin (Pola) was added to rituximab, ifosfamide, carboplatin, and etoposide (PolaR-ICE) as salvage therapy.
Time Frame: From initial treatment to the end of salvage therapy (up to three cycles).
Population: Three subjects were not evaluable for they did not finish two cycles of treatment.
Measure: Number (95% Confidence Interval); unit: percentage of ORR participants
Arm/Group | Treatment (PolaR-ICE)
Number analyzed (Participants) | 38
percentage of ORR participants | 83 [75 to 97]

ADVERSE EVENTS:
Time Frame: Averse events were assessed from the initial treatment to 30 days after the end of the treatment. Participants received three 21-day cycles of PolaR-ICE for salvage therapy and up to four 21-day cycles of Pola for consolidation therapy. Adverse events were monitored and assessed at each cycle treatment. Vital status was assessed from the initial treatment up to 2 years after the end of the treatment.
Arm/Group | Safety Lead-In | Phase II
All-Cause Mortality (participants affected / at risk) | 1/6 | 9/35
Serious Adverse Events (participants affected / at risk) | 1/6 | 8/35
Other Adverse Events (participants affected / at risk) | 6/6 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-In (N=6) | Phase II (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-In (N=6) | Phase II (N=35)
Anemia (Blood and lymphatic system disorders) | 6 (22) | 27 (86)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 5 (6)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 8 (15)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 4 (8)
Black stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2) | 2 (3)
Blood in stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (4) | 12 (18)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (6)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (7) | 22 (30)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (4) | 9 (10)
Chills (General disorders) | 0 (0) | 4 (4)
Covid positive (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 3 (3) | 3 (3)
Edema trunk (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 20 (27)
Fever (General disorders) | 1 (1) | 2 (2)
Injection site reaction (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 4 (4)
Bleeding gums (General disorders) | 0 (0) | 1 (1)
Petechiae (General disorders) | 0 (0) | 1 (1)
Rash (General disorders) | 0 (0) | 1 (1)
Eye infection (General disorders) | 0 (0) | 1 (1)
Folliculitis (General disorders) | 1 (1) | 0 (0)
Papulopustular rash (General disorders) | 0 (0) | 1 (1)
Tooth infection (General disorders) | 1 (1) | 2 (2)
Urinary tract infection (General disorders) | 0 (0) | 1 (1)
Vaginal infection (General disorders) | 0 (0) | 1 (1)
Furunculitis (General disorders) | 1 (1) | 0 (0)
Bruising (General disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 2 (2)
Infusion related reaction (General disorders) | 2 (2) | 4 (4)
Platelet Count Decreased (General disorders) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3) | 7 (11)
Alkaline phosphatase increased (Investigations) | 1 (1) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 6 (14)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 5 (6)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (2)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 1 (4) | 2 (3)
Lymphocyte count decreased (Investigations) | 6 (17) | 9 (17)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (5) | 20 (51)
Platelet count decreased (Investigations) | 6 (12) | 23 (87)
Weight gain (Investigations) | 1 (1) | 2 (3)
Weight loss (Investigations) | 3 (3) | 5 (10)
White blood cell decreased (Investigations) | 4 (7) | 18 (32)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 7 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 9 (17)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 6 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (7) | 7 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 6 (13)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5) | 9 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (4) | 8 (10)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
Dizziness (Nervous system disorders) | 1 (1) | 8 (9)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (4)
Headache (Nervous system disorders) | 1 (1) | 8 (13)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 12 (13)
Syncope (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 7 (8)
Dysuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Glucosuria (Renal and urinary disorders) | 0 (0) | 4 (4)
Hematuria (Renal and urinary disorders) | 1 (1) | 5 (5)
Proteinuria (Renal and urinary disorders) | 1 (1) | 4 (5)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vaginal itch (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 8 (11)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (3) | 12 (38)
Hypotension (Vascular disorders) | 1 (1) | 4 (4)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT04665765/Prot_SAP_000.pdf